CLINICAL TRIAL: NCT04097041
Title: Surgery Compared to Masking Device for Venous Pulsatile Tinnitus
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in availability of investigators/participants
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Peter Santa Maria, Assistant Professor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 43338
Record Dates: First submitted 2018-08-16; First posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Intervention Model Description: Surgery arm - patient undergoes tympanomastoidectomy (approx 2 hour operation on ear and mastoid) where a local soft tissue flap is transferred to cover the sigmoid sinus, a cartilage and perichondrial graft is taken from the tragus to cover the jugular bulb). Patient has routine follow up - H&P, 2 weeks after surgery and then H&P, Audiometry and Tympanometry over 12 months post surgery (3rd month, 6th month and 12th month). Non surgery arm - patient has audiological consult and fitting of masking device.
  The Patient has a routine follow up - H&P, 2 weeks after masking fitting and then H&P, Audiometry, Tympanometry over 12 months (3rd month, 6th month and 12th month). Patient cross over to change arms, at 6 months, if they have no resolution of symptoms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical Arm (Active Comparator): Surgery arm - patient undergoes tympanomastoidectomy (approx 2 hour operation on ear and mastoid) where a local soft tissue flap is transferred to cover the sigmoid sinus, a cartilage and perichondrial graft is taken from the tragus to cover the jugular bulb).Patient has routine follow up - H&P, 2 weeks after surgery and then H&P, Audiometry and Tympanometry over 12 months post surgery (3rd month, 6th month and 12th month).
  Interventions: Procedure: Tympanomastoidectomy
- Non-Surgery (Active Comparator): Non surgery arm - patient has audiological consult and fitting of masking device.
  The Patient has a routine follow up - H&P, 2 weeks after masking fitting and then H&P, Audiometry, Tympanometry over 12 months (3rd month, 6th month and 12th month). Patient cross over to change arms, at 6 months, if they have no resolution of symptoms.
  Interventions: Procedure: Tympanomastoidectomy; Procedure: Non-Surgery

INTERVENTIONS:
Procedure: Tympanomastoidectomy — Patient undergoes tympanomastoidectomy (approx 2 hour operation on ear and mastoid) where a local soft tissue flap is transferred to cover the sigmoid sinus, a cartilage and perichondrial graft is taken from the tragus to cover the jugular bulb).
Procedure: Non-Surgery — Screening performed at outpatient clinic after consultation for management of venous pulsatile tinnitus. Consent and formal recruitment into study performed at preoperative visit or at audiological visit.
  The masking device is a hearing aid that provides sound that is aimed to negate the internal sound from the pulsatile tinnitus. Almost all hearing aid can be converted to a masking device for tinnitus. It is externally worn on the ear and provides sound at a desired volume. The benefits of wearing the masking device are that it may reduce the volume of the pulsatile tinnitus. As it is worn on the external ear and is not invasive there are minimal risks but potential risks could include irritation of the external ear and discomfort from wearing.
  Arms: Non-Surgery

SUMMARY:
The investigators aim to study whether surgical resurfacing of the sigmoid sinus and jugular bulb will result in elimination of venous pulsatile tinnitus.

DETAILED DESCRIPTION:
Currently there is no known treatments with efficacy for venous pulsatile tinnitus without any pathology. The investigators hope to learn that in surgery, resurfacing of the sigmoid sinus and jugular bulb (acoustic dampening) will eliminate symptoms such as pulsatile tinnitus in patients. The knowledge learned will significantly help treat and alleviate future patients that have pulsatile tinnitus.

The purpose of the study is to examine whether surgical resurfacing of the sigmoid sinus and jugular bulb will result in elimination of pulsatile tinnitus in human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral venous pulsatile tinnitus
* Visual Analogue score of severity >5

Exclusion Criteria:

* Surgery exclusion criteria
* Only hearing ear
* Unfit for surgery / anesthesia
* Visual Analogue score of severity 5 or less

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-08 (Estimated); Primary Completion 2022-08-26 (Estimated); Study Completion 2023-08-26 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in patient-reported tinnitus score | 12 Months
  Tinnitus severity rated on a 10-point Likert scale (range: 1-10; higher scores correspond to more severe symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Santa Maria, MD, PhD, Principal Investigator — Stanford University

REFERENCES:
- [Result] Santa Maria PL. Sigmoid sinus dehiscence resurfacing as treatment for pulsatile tinnitus. J Laryngol Otol. 2013 Jul;127 Suppl 2:S57-9. doi: 10.1017/S0022215113000649. Epub 2013 Apr 18. PMID 23595093
- See also: Sigmoid sinus dehiscence resurfacing as treatment for pulsatile tinnitus. — https://www.ncbi.nlm.nih.gov/pubmed/23595093